CLINICAL TRIAL: NCT03945201
Title: Effect of a Virtual Reality-enhanced Exercise and Education Intervention on Patient Engagement and Learning in Cardiac Rehabilitation
Brief Title: Virtual Reality-enhanced Exercise and Education in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17P.652
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Adherence, Patient; Motivation; Satisfaction
Keywords: cardiac rehabilitation; virtual reality; VR; treadmill; education retention; patient education
MeSH Terms: conditions — Patient Compliance; Personal Satisfaction | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Consent and enrollment process does not mention virtual reality to maintain blinding between control and intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Participants receive normal cardiac rehabilitation according to approved standard of care. They use multiple pieces of exercise equipment at each session for increasing amounts of time and at incrementally increasing levels of difficulty. After establishing a baseline, participants are allowed to use the treadmill for "up to 15 minutes" at each session.
  Interventions: Other: Standard of care
- Virtual walking trails (Experimental): Participants use multiple pieces of exercise equipment at each session for increasing amounts of time and at incrementally increasing levels of difficulty. After establishing a baseline, participants are allowed to use the treadmill for "up to 15 minutes" at each session. The treadmill is positioned in front of a vertically oriented high definition television screen showing Bionautica Trails, virtual walking trails created by Plas.md.
  Interventions: Other: Virtual walking trails

INTERVENTIONS:
Other: Virtual walking trails — During time on the treadmill, participants walk in front of Bionautica Trails, the virtual walking trails created by Plas.md. Participants can select between seven trails including various nature themed trails and a space setting. While walking, participants wear wireless headphones that provide audio of cardiac rehabilitation education at random intervals. These education pieces cover six categories of information: Understanding Your Heart Condition, Diet, Exercise, Medication, Managing Risk Factors, and Emotional Health.
  Other Names: Bionautica Trails
  Arms: Virtual walking trails
Other: Standard of care — Participants receive normal standard of care cardiac rehabilitation, completing multiple pieces of exercise equipment at increasing intervals according to the Jefferson Methodist Cardiac Rehabilitation program's protocols. Participants are given the option to use the treadmill for "up to" 15 minutes.
  Arms: Standard of care

SUMMARY:
This study incorporates a virtual reality (VR) simulated walking environment, with audio component of patient education, into the treadmill portion of outpatient cardiac rehabilitation (CR). The VR program was developed by Plas.MD and is named Bionautica Trails.

ELIGIBILITY:
Inclusion Criteria:

* Participants must independently choose or be referred to Jefferson Health Methodist Cardiac Rehabilitation Program for outpatient cardiac rehabilitation.
* Participants must have a referring cardiac condition requiring cardiac rehabilitation therapy.

Exclusion Criteria:

* Physical inability to use treadmill
* Medically unsafe to use a treadmill for 15 minutes
* Inability to understand English
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Comparison of Participant 6-minute Walk Test Improvement Between Control and Intervention Groups | From date of enrollment through study completion, an average of 12 weeks
  Each participant will complete a 6MWT at both their first and last cardiac rehab treatment sessions. Distance improvement between first and last treatment session is expected for all participants. Average distance improvement (measured in feet) between study arms will be compared to evaluate effectiveness of interventions.

SECONDARY OUTCOMES:
Participant Satisfaction with Cardiac Rehab Treatment | At completion of cardiac rehab treatment, an average of 12 weeks
  All participants are asked to complete a satisfaction survey, utilizing likert scales and location specific questions to evaluate their satisfaction with treatment. Questions delineate the differences between experiences part of standard of care and those specific to the trial.
Participant Cardiac Education Retention | At enrollment; at date of treatment completion, average of 12 weeks; two months following treatment completion
  Participants will complete a brief, 5-question, education quiz at several times throughout their rehabilitation treatment. The quiz will be administered to establish a baseline of their cardiac knowledge prior to treatment, at the end of their treatment to evaluate primary comprehension, and again after treatment to evaluate longterm retention of information. Quiz scores and trends will be compared between study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson Health Methodist Cardiac Rehabilitation Program, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available for all gathered data, including primary and secondary outcomes, by request.
Supporting Information: Study Protocol
Time Frame: Data will be available by request indefinitely.
Access Criteria: Data will be available by request.

REFERENCES:
- [Background] Ades PA, Keteyian SJ, Wright JS, Hamm LF, Lui K, Newlin K, Shepard DS, Thomas RJ. Increasing Cardiac Rehabilitation Participation From 20% to 70%: A Road Map From the Million Hearts Cardiac Rehabilitation Collaborative. Mayo Clin Proc. 2017 Feb;92(2):234-242. doi: 10.1016/j.mayocp.2016.10.014. Epub 2016 Nov 15. PMID 27855953
- [Background] Davies P, Taylor F, Beswick A, Wise F, Moxham T, Rees K, Ebrahim S. Promoting patient uptake and adherence in cardiac rehabilitation. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007131. doi: 10.1002/14651858.CD007131.pub2. PMID 20614453
- [Background] Kerins M, McKee G, Bennett K. Contributing factors to patient non-attendance at and non-completion of Phase III cardiac rehabilitation. Eur J Cardiovasc Nurs. 2011 Mar;10(1):31-6. doi: 10.1016/j.ejcnurse.2010.03.006. Epub 2010 May 10. PMID 20457543
- [Background] Mikkelsen T, Korsgaard Thomsen K, Tchijevitch O. Non-attendance and drop-out in cardiac rehabilitation among patients with ischaemic heart disease. Dan Med J. 2014 Oct;61(10):A4919. PMID 25283618
- [Background] Vieira A, Gabriel J, Melo C, Machado J. Kinect system in home-based cardiovascular rehabilitation. Proc Inst Mech Eng H. 2017 Jan;231(1):40-47. doi: 10.1177/0954411916679201. Epub 2016 Dec 19. PMID 27913628
- [Background] Dithmer M, Rasmussen JO, Gronvall E, Spindler H, Hansen J, Nielsen G, Sorensen SB, Dinesen B. "The Heart Game": Using Gamification as Part of a Telerehabilitation Program for Heart Patients. Games Health J. 2016 Feb;5(1):27-33. doi: 10.1089/g4h.2015.0001. Epub 2015 Nov 18. PMID 26579590
- [Background] Lynggaard V, Nielsen CV, Zwisler AD, Taylor RS, May O. The patient education - Learning and Coping Strategies - improves adherence in cardiac rehabilitation (LC-REHAB): A randomised controlled trial. Int J Cardiol. 2017 Jun 1;236:65-70. doi: 10.1016/j.ijcard.2017.02.051. Epub 2017 Feb 21. PMID 28259552
- [Background] Dankner R, Drory Y, Geulayov G, Ziv A, Novikov I, Zlotnick AY, Moshkovitz Y, Elami A, Schwammenthal E, Goldbourt U. A controlled intervention to increase participation in cardiac rehabilitation. Eur J Prev Cardiol. 2015 Sep;22(9):1121-8. doi: 10.1177/2047487314548815. Epub 2014 Sep 2. PMID 25183694
- [Background] Shema SR, Brozgol M, Dorfman M, Maidan I, Sharaby-Yeshayahu L, Malik-Kozuch H, Wachsler Yannai O, Giladi N, Hausdorff JM, Mirelman A. Clinical experience using a 5-week treadmill training program with virtual reality to enhance gait in an ambulatory physical therapy service. Phys Ther. 2014 Sep;94(9):1319-26. doi: 10.2522/ptj.20130305. Epub 2014 May 1. PMID 24786944
- [Background] Sloot LH, van der Krogt MM, Harlaar J. Effects of adding a virtual reality environment to different modes of treadmill walking. Gait Posture. 2014 Mar;39(3):939-45. doi: 10.1016/j.gaitpost.2013.12.005. Epub 2013 Dec 18. PMID 24412269
- [Background] Meng K, Seekatz B, Haug G, Mosler G, Schwaab B, Worringen U, Faller H. Evaluation of a standardized patient education program for inpatient cardiac rehabilitation: impact on illness knowledge and self-management behaviors up to 1 year. Health Educ Res. 2014 Apr;29(2):235-46. doi: 10.1093/her/cyt107. Epub 2014 Jan 7. PMID 24399262
- [Derived] Gulick V, Graves D, Ames S, Krishnamani PP. Effect of a Virtual Reality-Enhanced Exercise and Education Intervention on Patient Engagement and Learning in Cardiac Rehabilitation: Randomized Controlled Trial. J Med Internet Res. 2021 Apr 15;23(4):e23882. doi: 10.2196/23882. PMID 33856355